CLINICAL TRIAL: NCT01600365
Title: "Prospective, Interventional, Randomized, Double-masked With the Use of Ganciclovir Gel 0.3% for Treatment of Conjunctivitis Caused by Adenovirus."
Brief Title: Evaluate the Use of Ganciclovir Gel 0.3% for the Treatment of Conjunctivitis Caused by Adenovirus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adapt Produtos Oftalmológicos Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADA-GAN-02/10
Record Dates: First submitted 2011-03-22; First posted 2012-05-17 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Conjunctivitis; Adenovirus.
Keywords: Conjunctivitis; adenovirus.
MeSH Terms: conditions — Conjunctivitis; Adenoviridae Infections | interventions — Lubricant Eye Drops; Ganciclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ganciclovir (Active Comparator): Ophthalmic gel ganciclovir 0,3%: applied in affected eye 4 times daily for 10 days
  Interventions: Drug: Ganciclovir
- Ophthalmic gel (placebo) (Placebo Comparator): ophthalmic gel (placebo)in the study eye
  Interventions: Drug: Ophthalmic gel (placebo)

INTERVENTIONS:
Drug: Ophthalmic gel (placebo) — Ophthalmic gel (placebo): applied in affected eye 4 times daily for 10 days
  Other Names: artificial tears
  Arms: Ophthalmic gel (placebo)
Drug: Ganciclovir — Ophthalmic gel ganciclovir 0,3%: applied in affected eye 4 times daily for 10 days
  Other Names: ganciclovir gel
  Arms: Ganciclovir

SUMMARY:
The purpose of this study is to study the use of ganciclovir gel 0.3% for treatment of conjunctivitis caused by adenovirus.

DETAILED DESCRIPTION:
To evaluate the efficacy and tolerability of ganciclovir ophthalmic gel for the treatment of conjunctivitis comparing to placebo (ophthalmic gel). Visual acuity test and slit lamp examination (biomicroscopy) will be performed at each visit to assess the signs/symptoms and the regression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with eye disease with a clinical diagnosis of adenovirus conjunctivitis.
* Patients of both gender aged over 18 years.
* Patients who are not pregnant or nursing.
* Patients able (legally and mentally) to understand and sign informed consent had been signed.

Exclusion Criteria:

* Patients who are in the presence of corticosteroids, either by topical ocular, periocular, intraocular or systemic, for less than 30 days of enrollment and who can not make a drug suspension.
* Patients with serious systemic diseases like AIDS, cancer, etc., which in the opinion of the investigator, may put the patient at risk.
* Patient with a single eye or vision in one eye.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
time to regression of the ocular symptomatology | 10 days
  Time to regression of ocular symptomatology compared to the baseline, as determined by clinical evaluation (biomicroscopy) performed on V1, V2 and V3, based on scale of absent, mild, moderate and severe.

SECONDARY OUTCOMES:
Development of sub-epithelial infiltrates | 10 days
  Development of sub-epithelial infiltrates,incidence for the study duration and severity at each follow-up visit (based on scale of absent, mild, moderate and severe)
Degree of Bulbar conjunctival Injection | 10 days
  Degree of bulbar conjunctival injection at each follow-up visit, based on the scale of mild, moderate and severe
Involvement of the second eye | 10 days
  Involvement of the second eye - incidence for the study duration and severity at each follow-up visit, as determined by the clinical evaluation (biomicroscopy)
Patient Dairy - intensity of ocular pain | 10 days
  intensity of ocular pain selected by the patient on the "Patient Dairy" based on the visual analogue scale (VAS)on each follow-up visit (absent, mild, moderate, severe)

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort, PhD, MD, Principal Investigator — Federal University of São Paulo